CLINICAL TRIAL: NCT00489346
Title: A Double-Blind, Randomized, Double-Dummy, Multicenter Study to Evaluate and Compare Oral Montelukast and Inhaled Fluticasone in the Control of Asthma for 6- to 14-Year-Olds With Mild Persistent Asthma
Brief Title: A Study to Evaluate MK0476 and Fluticasone to Control Asthma in Patients With Mild Persistent Asthma (0476-910)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-910; 2007_574
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Asthma, Bronchial
MeSH Terms: conditions — Asthma | interventions — montelukast; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0476, montelukast sodium / Duration of Treatment: 1 Year
Drug: Comparator : fluticasone propionate / Duration of Treatment: 1 Year

SUMMARY:
A study to evaluate MK0476 and Fluticasone to control asthma in patients with mild persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female, 6-14 years of age with mild persistent asthma
* Patient has a history of the following symptoms: wheezing, chest tightness, cough, etc.
* Patient has asthma diagnosed by a doctor

Exclusion Criteria:

* Patient is hospitalized
* Patient has had major surgery or participated in another clinical trial in the last 4 weeks
* Patient has been on a breathing tube for asthma

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 994 (Actual)
Dates: Start 2001-10; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Improvement of asthma with MK0476 and Fluticasone as measured by number of asthma rescue-free days | Duration of Trial

SECONDARY OUTCOMES:
Improved effect of MK0476 and fluticasone on FEV1 values | Duration of Trial

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Garcia Garcia ML, Wahn U, Gilles L, Swern A, Tozzi CA, Polos P. Montelukast, compared with fluticasone, for control of asthma among 6- to 14-year-old patients with mild asthma: the MOSAIC study. Pediatrics. 2005 Aug;116(2):360-9. doi: 10.1542/peds.2004-1172. PMID 16061590